CLINICAL TRIAL: NCT02375529
Title: Estudio Prospectivo Aleatorizado de la colecistectomía laparoscópica Por Puerto único vs colecistectomía laparoscópica Por Cuatro Puertos en Pacientes Con Colelitiasis sintomática y régimen de cirugía Sin Ingreso.
Brief Title: A Trial of Single Incision Versus Four Ports Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/19
Record Dates: First submitted 2014-11-12; First posted 2015-03-02 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2015-02

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Incision Cholesystectomy (SILC) (Experimental): Single Incision Laparoscopic Cholecystectomy (SILC): The umbilicus is grasped and a 2 cm vertical skin and fascial incision is performed. A multiport (TriPort®) is inserted under direct vision. Principles of cholecystectomy are the same as traditional laparoscopic cholecystectomy.
  Interventions: Procedure: Single Incision Laparoscopic Cholecystectomy (SILC)
- Four Ports Cholecystectomy (4PCL) (Active Comparator): Four Ports Conventional laparoscopic cholecystectomy (4PCL): A 10mm supraumbilical incision is made and the pneumoperitoneum insufflated through a Veress needle. 4 ports are introduced: 2 of 10mm in supraumbilical and left flank and 2 of 5mm in epigastric and right flank.
  Interventions: Procedure: Four Ports Laparoscopic Cholecystectomy (4PLC)

INTERVENTIONS:
Procedure: Single Incision Laparoscopic Cholecystectomy (SILC) — A 2.5-cm incision is made through the everted umbilicus down to the midline fascia, and through the fascia and the peritoneum. The multichannel port (Olympus) is introduced. Carbon dioxide is insufflated (12 mmHg) and a 30 degree 10-mm laparoscope is introduced. The operating table is put in the reverse Trendelenburg position (20 degrees), left side down. A pre-curved grasper and the monopolar electrocautery are introduced through the other 2 ports of the trocar and the dissection of the gallbladder starts in a retrograde manner. The triangle of Calot is exposed, the cystic duct and artery are separately dissected and ligated with 5 mm clips. The monopolar electrocautery is used to remove the gallbladder from the liver bed. The gallbladder is removed along with the port system from the abdominal cavity. The fascia at the port site is closed and the umbilicus is inverted.
  Arms: Single Incision Cholesystectomy (SILC)
Procedure: Four Ports Laparoscopic Cholecystectomy (4PLC) — An 11-mm periumbilical port, a 10-mm left upper quadrant port , 5mm subxyphoid port, and 5-mm right lower quadrant port were used in 4-port LC. We adopted the single surgeon technique in the 4-port LC using 30-degree operating telescopes that was inserted into the umbilical port. Retraction of the gallbladder was done by the long grasping forceps through the 5-mm right lower quadrant port, whereas dissection was accomplished through the 10-mm left upper quadrant port. The cystic duct and cystic artery were clipped by a 5-mm multiple clip applicator. The gallbladder was retrieved through the umbilical port after the position of the operating telescope was changed.
  Nontransparent surgical adhesive tape was applied to the standard 4-port sites at the end of the operation .
  Arms: Four Ports Cholecystectomy (4PCL)

SUMMARY:
Background: Single-incision laparoscopic cholecystectomy (SILC) is increasingly being used as a minimally invasive surgery with potential benefits over 4-port laparoscopic cholecystectomy (LC) in terms of postoperative pain and faster recovery.

Methods: Seventy-three patients with symptomatic cholelithiasis were randomized to SILC (n=37) or LC (n=36). Data measures included operative details, adverse events, postoperative pain and analgesic requirements, success of the ambulatory process, return to normal activity and return to work, cosmetic results and quality of life score.

ELIGIBILITY:
Inclusion Criteria:

* age higher than 18 and lower than 80
* American Society of Anesthesiologists class (ASA) I-II,
* absence of any previous anesthetic complication,
* accompaniment by a responsible adult during 24 hours,
* symptomatic gallstones candidate to cholecystectomy
* and a signed informed consent.

Exclusion Criteria:

* a Body Mass Index (BMI) higher than 35,
* any laparoscopic contraindication,
* acute cholecystitis background, suspect of Mirizzi's Syndrome, common duct stones or malignancy,
* anti-inflammatory allergy
* psychiatric history that could hinder ambulatory procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-05; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
evolution of postoperative pain | 2, 4, 6 and 8 postoperative hours, 1, 3, 7 and 30 days after surgery